CLINICAL TRIAL: NCT01974076
Title: A Study of Transcranial Direct Current Stimulation (tDCS) as an Adjunct to Cognitive Behavioural Therapy (CBT) for Depression
Brief Title: Transcranial Direct Current Stimulation (tDCS) as an Adjunct to Cognitive Behaviour Therapy (CBT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Belmont Private Hospital (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC13276
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Active Comparator)
  Interventions: Device: Active tDCS + CBT
- Sham tDCS (Sham Comparator)
  Interventions: Device: Sham tDCS + CBT

INTERVENTIONS:
Device: Active tDCS + CBT
  Arms: Active tDCS
Device: Sham tDCS + CBT
  Arms: Sham tDCS

SUMMARY:
This study will investigate whether transcranial direct current stimulation (tDCS) can enhance the efficacy of cognitive behavioural therapy for the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years old.
2. Have a DSM-IV diagnosis of Major Depressive Episode of minimum 4 weeks duration.
3. MADRS score ≥ 20 at study entry.

Exclusion Criteria:

1. Participant is unable to give informed consent.
2. DSM-IV diagnosis of psychotic disorder (lifetime).
3. Bipolar disorder diagnosis and not on a mood stabiliser.
4. Eating disorder (current or within past year).
5. Obsessive compulsive disorder (lifetime).
6. Post-traumatic stress disorder (current or within past year).
7. Mental retardation.
8. Drug or alcohol abuse or dependence (preceding 3 months).
9. Inadequate response to ECT (current episode of depression).
10. Rapid clinical response required, e.g., high suicide risk, inanition or psychosis.
11. Clinically defined neurological disorder or insult.
12. Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
13. Pregnancy.
14. Concurrent long acting benzodiazepines, ritalin or dexamphetamine medication.
15. Change in psychotropic medication during 2-week period prior to the study or during the course of the 3-week trial.
16. Participant becomes hypomanic or manic, as defined by DSM-IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 3 weeks

SECONDARY OUTCOMES:
Depression and Anxiety Stress Scale | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Belmont Private Hospital, Carina, Brisbane, Queensland, Australia